CLINICAL TRIAL: NCT00367497
Title: Phase 2 Study of Rituximab and ESHAP (Etoposide, Methylprednisolone, Cytarabine, and Cisplatin) in Relapsed and Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: Safety and Efficacy Study of Salvage Chemotherapy (R-ESHAP) to Treat Relapsed and Refractory Aggressive Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The stopping rule was applied because of low response rates.
Sponsor: Keio University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-40
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: aggressive non-Hodgkin's lymphoma; salvage chemotherapy; rituximab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Etoposide; Methylprednisolone; Cytarabine; Cisplatin

INTERVENTIONS:
Drug: Rituximab, Etoposide, Methylprednisolone, Cytarabine, Cisplatin

SUMMARY:
Aggressive non-Hodgkin's lymphoma is difficult to handle once it relapses or becomes refractory to chemotherapy. Various second or third line chemotherapies, which are called salvage chemotherapy, were developed without promising results. Improvement in efficacy by adding relatively new agent, rituximab, to chemotherapy is now widely accepted in non-Hodgkin's lymphoma. This study will test the safety and efficacy of adding rituximab to existing salvage chemotherapy, ESHAP (R-ESHAP). Our aim is also to proceed to high-dose chemotherapy with autologous hematopoietic stem cell transplantation after successful R-ESHAP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of aggressive non-Hodgkin's lymphoma
* Refractory to the first line chemotherapy or relapsed
* Expression of CD20 on lymphoma cells
* Measurable lesions on imaging studies

Exclusion Criteria:

* Blood cell counts not reaching to 3,000/microliter for white blood cells, 7 g/dl for hemoglobin, and 50,000/microliter for platelets without transfusion at the time of registration
* Circulating lymphoma cells equal to or more than 25,000/microliter
* Hepatic dysfunction
* Renal insufficiency
* Cardiac dysfunction or arrhythmia
* Sever infection (bacterial, viral)
* CNS involvement
* Other malignancies
* Pregnancy or breast feeding

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-08; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Overall response

SECONDARY OUTCOMES:
Complete response
Safety
Overall survival
Progression free survival
Effectiveness of peripheral blood stem cell collection

CONTACTS AND LOCATIONS:
Overall Officials: Norihiro Awaya, MD, PhD, Principal Investigator — Keio University
Locations (1):
- Keio University School of Medicine, Tokyo, Japan